CLINICAL TRIAL: NCT06732128
Title: Nature-based Virtual Reality Intervention for Depression in Alzheimer's Disease: a Pilot Randomized Controlled Trial
Brief Title: Nature-based Virtual Reality Intervention for Depression in Alzheimer's Disease
Acronym: VRN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: St. Mary's Research Center, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VRN
Record Dates: First submitted 2024-11-19; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Alzheimer Disease; Depression
Keywords: virtual reality
MeSH Terms: conditions — Alzheimer Disease; Depression | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Participants will receive nature-based applications available on the Oculus platform, as well as nature-based 360 videos with the same content as the control group however in a 360 format.
  Interventions: Other: nature-based virtual reality applications and videos
- Control Group (Active Comparator): Participants will receive YouTube links to watch nature-based videos on a device (e.g., a tablet).
  Interventions: Other: nature-based videos

INTERVENTIONS:
Other: nature-based virtual reality applications and videos — Participants will receive nature-based applications available on the Oculus platform, as well as nature-based 360 videos with the same content as the control group however in a 360 format.
  Arms: Treatment Group
Other: nature-based videos — Participants will receive YouTube links to watch nature-based videos on a device (e.g., a tablet).
  Arms: Control Group

SUMMARY:
Behavioural and psychological symptoms of dementia (BPSD), such as depression affect up to 90% patients with dementia. Non-pharmacological treatment of BPSD, can be difficult to access, require caregiver support, travel, and often have long waiting lists. Virtual reality (VR) is an innovative, portable, immersive, and accessible technology which can be used in-home. More information is required on the feasibility of using VR in-home with older adults with dementia.

Our study will offer a 4-week program of 15-minutes sessions, twice per week nature-based VR program for BPSD delivered in-home by virtual reality (VR). Additionally, caregivers will have the option of taking part in the study and provide feedback regarding the VR intervention. If successful, this project has the potential to prolong aging in place for individuals with BPSD, as BPSD is a significant factor in institutionalization.

DETAILED DESCRIPTION:
The burden of dementia is rapidly growing, affecting nearly 50 million individuals globally and costing $818 billion dollars yearly. Alzheimer's disease (AD) is the most common form of dementia. AD includes changes in mood and behavior, referred to as the behavioral and psychological symptoms of dementia (BPSD). Depression is among the most common BPSD, impacting 50% of older adults with AD. Existing pharmacological treatment for depressive symptoms in AD (AD-D) lack evidence for efficacy and have many potential side effects (e.g. cognitive impairments, falls, mortality), Non-pharmacological interventions have been recommended but are associated with significant challenges such as travel, cost and the difficulty in accessing specialized therapists.

Virtual reality (VR), an immersive audiovisual technology, can address these challenges as it is an accessible and cost-effective intervention which can be delivered in a variety of settings. VR can easily be delivered in-home, and therefore address many of the limitations of traditionally delivered non-pharmacological interventions, such as accessibility, intervention non-adherence and difficulties with maintaining intervention frequency. Additional technology will be utilized to collect physiological data such as movement using the Fitbit Charge 6 and a Muse headband will measure electroencephalogram (EEG). Previous literature on VR based intervention for older adults is limited, with very few randomized control trials, rather it is primarily case studies, cross-sectional studies, and non-immersive VR. However, there are no studies assessing in-home VR for individuals with AD or for AD-D.

We propose a pilot randomized controlled trial (RCT) to assess nature-based VR intervention (N-VR) for AD-D. We will randomize (1:1) 50 participants with AD-D to N-VR vs. an active control intervention of various nature-based videos (N-CI). All participants will receive the intervention as 15-min sessions delivered twice a week, assessor-blinded, for 4 weeks. Assessments will be conducted at baseline, within 7 days of starting the intervention, at follow-up, within 7 days of completing the 4-week course, and after each 15-min session.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild to early-moderate stage AD (including mixed dementia with AD) using the Diagnostic and Statistical Manual of Mental Disorders, 5th Ed. Criteria
* Age of 50 years or older
* Medical stability to participate in the trial
* Patient Health Questionnaire score 5-14
* Investigator judgement on whether the participant is comfortable with technology
* Access to WiFi and a smart device for connecting on WebEx and downloading the Fitbit and Muse applications
* Have someone available to be present during all sessions

Exclusion Criteria:

* Unstable medical or psychiatric condition, including substance use based on an investigator opinion
* Visual or hearing impairments that would impair participation
* Patient Health Questionnaire score 15-27 and/or score of 1 or 2 in section E question 1 of the Cornell Scale for Depression in Dementia
* Any other reason, which will make the study participation intolerable for the participant in the opinion of the study investigator

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2025-06-11 (Estimated); Study Completion 2025-11-11 (Estimated)

PRIMARY OUTCOMES:
Tolerability of nature-based virtual reality | 4 weeks
  Hypothesis 1a (Tolerability): Using the Simulator Sickness Questionnaire (SSQ) at the end of the last session, the mean SSQ score for N-VR group will be less than 10 (with 10 or more being the cut-off for clinically significant cybersickness)
Feasibility of nature-based virtual reality | 4 weeks
  The number of sessions completed and major/minor technical issues during the session.
Acceptability of nature-based virtual reality | 4 weeks
  The Personal Involvement Inventory (PII) score mean after the last N-VR completed session.

SECONDARY OUTCOMES:
Depression in AD-D | 4 weeks
  The Cornell Scale for Depression in Dementia (CSDD) score improvement over 4 weeks for the N-VR versus control group.

OTHER OUTCOMES:
Caregiver participant exploratory outcome | 4 weeks
  The experiences of AD-D participants' caregivers with the VR intervention, VR usability with AD-D, what they liked/had challenges with, and feedback for future VR use with this population (qualitative-focus group).
AD-D participant exploratory outcome - quality of life | 4 weeks
  The preliminary efficacy of N-VR in improving quality of life in individuals with AD-D using the Quality of Life in Alzheimer's Disease (QOL-AD).
AD-D participant exploratory outcome - perceived stress | 4 weeks
  The preliminary efficacy of N-VR in improving stress in individuals with AD-D using the Perceived Stress Scale (PSS) and data from the Fitbit Charge 6.
AD-D participant exploratory outcome - attention | 4 weeks
  The preliminary efficacy of N-VR in improving attention in individuals with AD-D using the Montreal Cognitive Assessment (MoCA) attention task.
AD-D participant exploratory outcome - pleasure | 4 weeks
  The preliminary efficacy of N-VR in improving pleasure in individuals with AD-D using the Snaith-Hamilton Pleasure Scale (SHAPS).
AD-D participant exploratory outcome - sleep | 4 weeks
  The preliminary efficacy of N-VR in improving sleep in individuals with AD-D determined by the number of hours the participant slept, collected by the Fitbit Charge 6.
AD-D exploratory outcome - calmness | 4 weeks
  The preliminary efficacy of N-VR in improving calmness in individuals with AD-D using data from the Muse headband.
AD-D exploratory outcome - loneliness | 4 weeks
  The preliminary efficacy of N-VR in decreasing loneliness in individuals with AD-D using the UCLA loneliness scale.
AD-D exploratory outcome - nature relatedness | 4 weeks
  The preliminary efficacy of N-VR in improving nature relatedness in individuals with AD-D using the Nature-Relatedness Scale short version (NR-6).
AD-D participants exploratory outcome - activity | 4 weeks
  The preliminary efficacy of N-VR in increasing activity in individuals with AD-D, determined by baseline vs post-assessment average over 5 days using Fitbit.
AD-D participant exploratory outcome - presence | 4 weeks
  The preliminary efficacy of N-VR in improving presence in individuals with AD-D using the Slater-Usoh-Steed Presence Questionnaire (SUS).
AD-D participant exploratory outcome - immersion | 4 weeks
  The preliminary efficacy of N-VR in improving immersion using the Immersive Tendencies Questionnaire (ITQ).

CONTACTS AND LOCATIONS:
Overall Officials: HARMEHR SEKHON, PhD, Principal Investigator — CAMH and McGill/St. Mary's Research Centre; Eric Brown, MD, Principal Investigator — CAMH and UofT
Locations (1):
- Centre for Addictions and Mental Health (CAMH), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No